CLINICAL TRIAL: NCT03931824
Title: Efficacy Of Platelet Rich Plasma In The Treatment Of Hemiplegıc Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Hale Karapolat, Professor in Physical Medicine and Rehabilitation Department, Ege University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRP-HSP
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Shoulder Pain; Shoulder Impingement; Hemiplegia, Infantile; Shoulder Subluxation; Spasticity, Muscle
Keywords: Shoulder Pain; Hemiplegia; Shoulder Subluxation; Spasticity; Stroke
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome; Hemiplegia; Muscle Spasticity; Stroke | interventions — Exercise; Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Solutions were prepared by an investigator, and injectors were coated with an opaque layer in order to conceal the content from both the one performing the injection and the patients. Data was then analyzed by an investigator who was blind to the study groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP group (Experimental): A venous blood sample of 8.5 ml were obtained from patients. For the study group, the blood samples were mixed with 1.5 ml ACD-A or sodium citrate to achieve anticoagulation. Resulting material was then centrifugated for 5 minutes with RCF 1200 G speed to clump erythrocytes, and then centrifugated for 10 minutes in same speed to obtain thrombocyte concentrate. 2 ml's of the platelet rich plasma was injected to the shoulder of the subjects. For the sham injection group, same amount of blood was taken and they were given a of waiting time of same duration with the study group, with the resulting preparate being 2 ml's of 0,9% saline instead. PRP solutions were prepared with kits of Easy PRP(Neotec Biotechnology, Istanbul, Turkey).
  Injections were done every two weeks, for a total of 3 times.
  Interventions: Other: PRP; Other: Exercise
- Placebo group (Sham Comparator): Injections containing saline were done every two weeks, for a total of 3 times. 21 G injection needles with injection technique of posterior approach were used. To provide blindness, all injections were done using injectors coated with non transparent tape. All of the PRP injections were done by the same physician each time, with compliance to preventive measures against complications such as infections. Patients and the physician who applied the injection were blinded to the groups, and the solution was prepared by another researcher who was not blind to the groups.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: PRP — A venous blood sample of 8.5 ml were obtained from patients. For the study group, the blood samples were mixed with 1.5 ml ACD-A or sodium citrate to achieve anticoagulation. Resulting material was then centrifugated for 5 minutes with RCF 1200 G speed to clump erythrocytes, and then centrifugated for 10 minutes in same speed to obtain thrombocyte concentrate. 2 ml's of the platelet rich plasma was injected to the shoulder of the subjects. For the sham injection group, same amount of blood was taken and they were given a of waiting time of same duration with the study group, with the resulting preparate being 2 ml's of 0,9% saline instead. PRP solutions were prepared with kits of Easy PRP(Neotec Biotechnology, Istanbul, Turkey).
  Injections were done every two weeks, for a total of 3 times. 21 G injection needles with injection technique of posterior approach were used(18, 19). To provide blindness, all injections were done using injectors coated with non transparent tape.
  Other Names: Platelet rich plasma injections
  Arms: PRP group
Other: Exercise — All of the patients were also informed about proper positioning and the standard care for the affected extremity. Their process of neurological rehabilitation was not changed, which was 5 days of the week, one session of 45 minutes a day. They were also given a program of standardized ROM exercises, which included passive and active motions.
  Other Names: Rehabilitation

SUMMARY:
In this study assessing whether platelet rich plasma injections(PRP) are effective in the management hemiplegic shoulder pain, 55 patients with hemiplegic shoulder pain was recruited to this randomized controlled study. Patients were randomized into two groups, first getting PRP injections, and other group taking sham injections.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were being an adult stroke patient with more than two weeks of shoulder pain and restriction, and not having a history of stroke before the recent incident.

Exclusion Criteria:

* Patients with aphasia, severe cognitive or psychiatric disorders, history of trauma, recent injection (<3 months) or surgery on the affected joint, complex regional pain syndrome, infections, pregnancy, thrombocytopenia(<150000 per microliter) or coagulation disorders or severe spasticity of the affected limb(Modified Ashworth Scale >3) were excluded from the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-01-07 (Actual); Primary Completion 2015-11-18 (Actual); Study Completion 2015-11-18 (Actual)

PRIMARY OUTCOMES:
Visual Analogous Scale | 3 months
  Visual Analogous Scales for pain were used as outcome measures. Both resting and activity pain levels were evaluated. Patients were asked to describe their pain, level of disability or treatment satisfaction on a 10 cm long line, with 0 point being "none", and 10 cm point being "highest possible". The proximity of the marked point to the 0 end was measured, and the results were recorded

SECONDARY OUTCOMES:
Shoulder ranges of motion | 3 months
  Shoulder range of motions were also evaluated as outcome measures. The measurements were done accordingly to the guidelines of American College of Orthopedic Surgeons by a conventional goniometer(20, 21). The researcher who performed the measurements was an experienced in this field, and was blinded to the treatment groups. External and internal rotation, adduction, abduction, flexion and extension of both shoulders were recorded for each group.
Functional Independence Measure(FIM) | 3 months
  Functional Independence Measure(FIM) is used to evaluate independence for the activities of daily living. It was developed to measure the results of the rehabilitation on the patient, and Turkish version of the tool shown to be valid and reliable in 2001. Having motor and cognitive subscales, the higher scores in FIM are interpreted as better functional independence.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege university school of medicine, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Uzdu A, Kirazli Y, Karapolat H, Unlu B, Tanigor G, Calis FA. Efficacy of platelet-rich plasma in the treatment of hemiplegic shoulder pain. Neurol Sci. 2021 May;42(5):1977-1986. doi: 10.1007/s10072-020-04710-0. Epub 2020 Sep 29. PMID 32990858